CLINICAL TRIAL: NCT01643057
Title: Stochastic Resonance Mattress (Physiological Interventions) and Biomarkers for Enhancing Neonatal Health
Status: Completed | Type: Observational
Sponsor: Wyss Institute at Harvard University (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Other Study IDs: AMD-CS-0015
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Apnea of Prematurity
Keywords: Apnea; Prematurity; Biomarkers; Stochastic Resonance; Neonatal
MeSH Terms: conditions — Apnea; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stochastic Resonance Mattress: The infant's isolette mattress will be replaced with a specially designed mattress (non-commercially available, designed by engineers at the Wyss Institute, Harvard University) to provide gentle vibrations and sounds during mattress stimulations.
  Interventions: Device: Stochastic Resonance Mattress

INTERVENTIONS:
Device: Stochastic Resonance Mattress — The infant's isolette mattress will be replaced with a specially designed mattress (non-commercially available, designed by engineers at the Wyss Institute, Harvard University) to provide gentle vibrations and sounds during mattress stimulations.

SUMMARY:
The purpose of this study is to explore physiological interventions and biomarkers for Apnea of Prematurity in newborn infants.

DETAILED DESCRIPTION:
Apnea of prematurity is defined as cessation of breathing that lasts for more than 20 seconds and/or is accompanied by oxygen desaturation or a decrease in heart rate (bradycardia). Because apnea presents itself within a variety of diseases in newborns, its diagnosis is based largely on the exclusion of other findings. The difficulty in relating the manifestation of apnea to its cause can lead to issues regarding appropriate medical management and delays in treatment.

Our exploration of physiological interventions for Apnea of Prematurity begins with stochastic resonance. Stochastic resonance is the introduction of noise to a system, to alter the system's behavior. This technology has been examined in previous medical applications. The hypothesis for this work is that stochastic resonance stimulation, in the form of gentle vibrations, will stabilize immature breathing patterns in infants.

In this research study, we will use an apnea mattress developed by engineers at the Wyss Institute, Harvard University, which provides gentle vibrations to the infant. We will closely follow the research protocol from UMass Medical School. Whilst the infant is on the mattress, clinical care data will be collected to determine effect on breathing patterns. We also hope to collect enough baseline and intervention data signals to be able to identify candidate biomarkers for apnea. This will assist in development of predictive algorithms for apnea in infants.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects are infants currently inpatient in the NICU at Beth Israel Deaconess Medical Center and:

* Born premature, at a gestational age < 36 weeks
* Demonstrate irregular breathing by having had at least one documented clinical apnea (> 20 seconds), bradycardia (< 100 bpm) and/or desaturation (< 90%)

Exclusion Criteria:

Eligible infants meeting the inclusion criteria above will be excluded from participation in the study if he/she:

* Is at a Post Conceptual Age of > 45 weeks at time of study (Calculated as: weeks of age at birth + weeks of age since birth)
* Has demonstrable pulmonary disease at time of study, i.e. Chronic Lung Disease, Infant Respiratory Distress Syndrome
* Has Hypoxic-Ischemic Encephalopathy including a cord pH of ≤ 7
* Has a congenital abnormality
* Has a genetic syndrome
* Has an anatomic brain anomaly
* Has hydrocephalus or intraventricular hemorrhage > Grade 3 or 4
* Is anemic (hemoglobin < 8g/dL)
* Has an infection at time of study
* Is undergoing therapeutic hypothermia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants currently inpatient in the Neonatal Intensive Care Unit at Beth Israel Deaconess Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Investigate effects of mattress intervention on breathing patterns | Each study session may last up to 24 hours. Participants may take part in up to 4 study sessions.
  Focus on inter-breath intervals and oxygen desaturation.

SECONDARY OUTCOMES:
Candidate Biomarkers for Apnea of Prematurity | Each study session may last up to 24 hours. Participants may take part in up to 4 study sessions.
  Candidate biomarkers in cardio-pulmonary, temperature, audiometry, photometry and clinical assessment data.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent C Smith, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center; David Paydarfar, MD, Principal Investigator — UMASS Medical School
Locations (1):
- Beth Israel Deaconness Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Smith VC, Kelty-Stephen D, Qureshi Ahmad M, Mao W, Cakert K, Osborne J, Paydarfar D. Stochastic Resonance Effects on Apnea, Bradycardia, and Oxygenation: A Randomized Controlled Trial. Pediatrics. 2015 Dec;136(6):e1561-8. doi: 10.1542/peds.2015-1334. PMID 26598451